CLINICAL TRIAL: NCT03360162
Title: Velocimetric Study of Temporal Arteries in Patients With Horton Disease Using Scan-Doppler
Acronym: VELHOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: VELHOR ( 29BRC17.0227)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Horton Disease
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of ultrasonography in detecting giant cell arteritis ( GCA) is emerging. Currently, temporal biopsy is the gold standard to diagnose GCA but studies have shown the interest to use B mode ultrasonography. However, until now, the study of velocities in GCA have not been yet performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspicious giant arteritis

Exclusion Criteria:

* patients who have already been treated or diagnosed for giant arteritis

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients aged more than 55 years old who are suspected of giant arteritis
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Velocimetric Study of Temporal Arteries in Patients With Horton Disease Using Scan-Doppler | 2 months
  velocimetric temporal arterial study in giant arteritis

SECONDARY OUTCOMES:
evaluation of the halo sign in giant arteritis using B mode ultrasonography | 2 months
  presence or absence of the halo sign in giant arteritis patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France